CLINICAL TRIAL: NCT01330082
Title: Efficacy of Adjunctive Photodynamic Therapy Using Light-emitting Diode in the Treatment of Chronic Periodontitis
Brief Title: Adjunctive Photodynamic Therapy in the Treatment of Chronic Periodontitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Tehran University of Medical Sciences, Tehran University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09123209916
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Periodontitis
Keywords: Photodynamic therapy; Light-emitting diode; toluidine blue; scaling and root planing
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Photodynamic therapy (Experimental): will be treated by PDT using Light-emitting diod(LED) (625-635nm,200mw/cm2 ,30 s for each site, fotoson CMS Dental ,Denmark) in the presence of toluidine blue O (TBO)
  Interventions: Other: Adjunctive Photodynamic Therapy
- Light-emitting diode Irradiation (Experimental): will be treated only by using Light-emitting diode(LED) (625-635nm,200mw/cm2 ,30 s for each site, fotoson CMS Dental ,Denmark)
  Interventions: Other: Light-emitting diod Irradiation
- applying photosensitizer (Experimental): will be treated only by toluidine blue O
  Interventions: Other: applying Photosensitizer

INTERVENTIONS:
Other: Adjunctive Photodynamic Therapy — using Light-emitting diod(LED) (625-635nm,200mw/cm2 ,30 s for each site, fotoson CMS Dental ,Denmark) in the presence of toluidine blue O (TBO)
  Arms: Photodynamic therapy
Other: Light-emitting diod Irradiation — 625-635nm,200mw/cm2 ,30 s for each site, fotoson CMS Dental ,Denmark
  Arms: Light-emitting diode Irradiation
Other: applying Photosensitizer — toluidine blue O is applied at the bottom of each periodontal pocket
  Arms: applying photosensitizer

SUMMARY:
The aim of this randomized clinical trial is to clinically evaluate the effectiveness of the adjunctive use of photodynamic therapy (PDT) with an light-emitting diode (LED) light source in the treatment of chronic periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. clinically diagnosis of advanced chronic periodontitis with more than 3 mm clinical attachment loss
2. presence of at least two teeth with probing depth of 4 to 6 mm without furcation involvement in each quadrant
3. at least 16 remaining teeth
4. no periodontal treatment in the past 12 months
5. no evidence of systemic disease related to periodontal problems
6. no use of antibiotics for the past 6 months
7. No smoking more than 10 cigarettes per day
8. no addiction to any kind of drugs
9. no pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline, one month, three month
  distance from gingival margin to base of the clinical pocket by William's periodontal probe

SECONDARY OUTCOMES:
Clinical attachment loss | Baseline, one month, three month
  distance in millimeter from a fix reference point (cement-enamel junction) to the bottom of probable pocket at experimental sites
Bleeding upon probing | Baseline, one month, three month
  presence or the absence of bleeding up to 30 second after probing with a William's periodontal probe
plaque index | Baseline,before PDT procedure, one month, three month
  teeth number 16,12,24,36,32,44 are evaluated according to silness plaque index instruction were scored between 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Neda Moslemi, DDS,MS, Study Chair — Tehran University of Medical Sciences; Seyed Hossein Bassir, DDS, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran